CLINICAL TRIAL: NCT07106164
Title: The Effect of Total Body Massage on Neonatal Jaundice in Preterm Neonates: A Randomized Controlled Trial
Brief Title: The Effect of Total Body Massage on Neonatal Jaundice in Preterm Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mariam Ibrahim, assistant professor of pediatrics and neonatology , Ain Shams University, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: total body massage & jaundice
Record Dates: First submitted 2025-07-17; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Preterm; Neonatal Hyperbilirubinemia
MeSH Terms: conditions — Premature Birth; Hyperbilirubinemia, Neonatal

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- total body massage (Experimental): patients received total body massage and phototherapy
  Interventions: Procedure: total body massage; Device: photo therapy
- control (Active Comparator): neonates received phototherapy only
  Interventions: Device: photo therapy

INTERVENTIONS:
Procedure: total body massage — Massage was done using the Field's Technique after starting phototherapy till discontinuation of phototherapy for 15 - 20 minutes, three times daily 1 hour after the morning, mid- day feeds and at night.
  Arms: total body massage
Device: photo therapy — neonates received phototherapy for the neonatal hyperbilirubinemia

SUMMARY:
Different methods are subscribed for the lowering of the bilirubin level, the most important of which are: exchange transfusion, phototherapy and using pharmacological agents. However, the remedial practice that has become most common for curing hyperbilirubinemia is phototherapy, has several side-effects. Thus there is constant research going on to find a substitute for phototherapy or to lessen its duration such as total body massage.

DETAILED DESCRIPTION:
Neonatal jaundice or hyperbilirubinemia is mostly cured (20% cases) though it can still prove hazardous and need medical intervention The most life-threatening case arising from this condition is kernicterus. Unfortunately, this condition is fatal in 75% cases and 80% of those who stay alive do not escape unscathed and exhibit problems related to the nervous system. Thus a timely cure of neonatal hyperbilirubinemia has become a major preventive measure Different methods are subscribed for the lowering of the bilirubin level, the most important of which are: exchange transfusion, phototherapy and using pharmacological agents . However, the most used treatment for curing hyperbilirubinemia is phototherapy, which has several side-effects ranging from doing harm to the cornea and the genital region to causing dehydration, diarrhoea and bronze kid syndrome. Thus there is constant research going on to find a substitute for phototherapy or to lessen the duration of the same.

Infant massage is a traditional practice in several regions of the world, to be more precise, in the cultures of Africa and Asia. A survey done recently in Bangladesh showed that 96% of the caretakers of neonates engaged in massaging the whole body of the infant one to three times a day. Healthcare practitioners in the West have also started to show interest in infant massage, especially, as an interventional measure for infants in neonatal intensive care units (NICUs) where mostly the environment is stressful and lacks adequate tactile stimulation. In order to promote infant growth, more parents and caretakers of low-risk babies are being trained in massage in the Western world studies have showed that massage stimulation encourages the passing of more meconium containing bilirubin by newborns and suggested that neonate massage can contribute toward the prevention of neonatal jaundice and the controlling of bilirubin to within normal range Taking all the above into account, this research was carried out with the aim of studying the effect of massage, using Field's Technique, on neonatal jaundice in preterm newborns on phototherapy.

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonates from 32 to 36 wks gestational age.
* Hyperbilirubinemia needing phototherapy.

Exclusion Criteria:

* Serious congenital malformation.
* Fetal hydrops.
* Hemolytic jaundice.
* Confirmed intrauterine infection (toxoplasmosis, rubella, cytomegalovirus, syphilis and herpes).
* Bilirubin level near exchange transfusion level.
* Any skeletal abnormality or joint affection.

Ages: 1 Hour to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
stool motions per day | baseline and daily throughout study completion, an average of 3 months
  Number of times the newborn passes stool will be recorded daily throughout phototherapy and total body massage
bilirubin level | baseline and throughout study completion, an average of 3 month
  Serum bilirubin recorded on the start of treatment before any massage intervention and regular follow up till discontinuation of phototherapy and rebound level upon stoppage of phototherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Childrens Hospital Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
data can be shared upon reasonable request from the corresponding author
Supporting Information: Study Protocol, SAP
Time Frame: after publication